CLINICAL TRIAL: NCT02249806
Title: Zürich Pulmonary Hypertension Outcome Assessment Cohort
Acronym: ZHPHCohort
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: 2014-0214_ZH PH Cohort
Record Dates: First submitted 2014-09-16; First posted 2014-09-26 (Estimated); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: Pulmonary Hypertension Outcome Assessment
Keywords: Pulmonary Hypertension; Chronic thromboembolic pulmonary hypertension; Pulmonary arterial hypertension; Outcome
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Arterial Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples Without DNA — Venous blood will be collected for serum markers and micro-RNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PH target therapy: Patients receiving PH target therapy
  Interventions: Other: PH target therapy according to physician

INTERVENTIONS:
Other: PH target therapy according to physician — Patients receiving PH target therapy

SUMMARY:
PH is a serious disease with a dismal prognosis and impaired quality of life when left untreated. Reliable patient centered and prognostically relevant outcome measures are highly warranted in the field of PH. With this prospective cohort study the investigators intend to gain important information on the course of the disease and knowledge on the value of different new and already established outcome parameters.

DETAILED DESCRIPTION:
PH is a serious disease with a dismal prognosis and impaired quality of life when left untreated. Advances in medical therapy have improved survival according to recent registries, but are associated with high healthcare costs. Most treatment trials and clinical follow-up assessments rely on the 6 minute walk distance as main outcome parameter although submaximal exercise performance reflects only one disease aspect.

Reliable patient centered and prognostically relevant outcome measures are highly warranted in the field of PH. With this prospective cohort study the investigator intend to gain important information on the course of the disease and knowledge on the value of different new and already established outcome parameters. New outcomes to be assessed will be home based activity monitoring, novel physiological measures, namely cerebral and muscle tissue oxygenation at rest and during exercise testing, stair ascent on mechanograph, sit to stand test and several serum markers and micro-RNA. All these assessments will be compared with hard endpoints events (death, lung-transplantation, hospitalization for PH), and with traditional outcome measures such as NYHA functional class, 6 minute walk distance, generic quality of life, cardiopulmonary exercise tests, sleep studies, health preference (utility) and cognitive function.

ELIGIBILITY:
Inclusion Criteria:

* Patients with precapillary pulmonary hypertension
* Adult male and female patients of all ages referred to our center for evaluation/treatment of PH
* Written informed consent by the subject after information about the research project

Exclusion Criteria:

* Patients with severe concomitant left heart disease (left ventricular ejection fraction <40%).
* Patients with restrictive lung disease (FVC<60% predicted); obstructive lung disease (forced expiratory volume (FEV) <60% predicted, with FEV 1/FVC<70%).
* Patients with any other disease limiting their ability to move (skeletal disease, neurological disease, etc.)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with precapillary pulmonary hypertension classified according to WHO
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-09; Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Survival | 10 years
  Transplant free survival will be registered
Change in the 6 minute walk distance | 10 years
  The change in 6 minute walk distance will be registered at 3, 6, 12 months and yearly thereafter

SECONDARY OUTCOMES:
New York Heart association (NYHA) functional class | 10 years
  The change in NYHA class will be registered at 3, 6, 12 months and yearly thereafter
Score in health related Quality of Life (HRQoL) questionnaires | 10 years
  The change in HRQoL class will be registered at 3, 6, 12 months and yearly thereafter
Hemodynamic parameters by echocardiography | 10 years
  The change in echo parameters will be registered at 3, 6, 12 months and yearly thereafter
Hospital days | 10 years
  Days spent in the hospital
red- and white blood cell counts | 10 years
  The change in blood cell count will be registered at 3, 6, 12 months and yearly thereafter
Partial pressures of oxygen and carbon dioxide, pH, bicarbonate, electrolytes | 10 years
  The change in arterial blood gas parameters taken from radial artery will be registered at 3, 6, 12 months and yearly thereafter, (ABL '90Flex'-blood gas analyzer, Radiometer, Switzerland)
Score on Short-Form-6 D, Euro-Qol 5 D (EQ-5 D), visual analogue scale, time trade-off, standard gamble test | 10 years
  The change in utility will be registered at 3, 6, 12 months and yearly thereafter
Overnight sleep study parameters | 10 years
  The change Overnight sleep study parameters will be registered at 3, 6, 12 months and yearly thereafter
Score in cognitive function tests | 10 years
  The change cognitive function will be registered at 3, 6, 12 months and yearly thereafter
Cardiopulmonary exercise test parameters | 10 years
  The change cardiopulmonary exercise test parameters will be registered at 3, 6, 12 months and yearly thereafter
ECG parameters | 10 years
  The change in ECG parameters will be registered at 3, 6, 12 months and yearly thereafter
Motion, step counts, metabolic equivalent | 10 years
  The change in Activity assessment parameters will be registered at 3, 6, 12 months and yearly thereafter with actigraphy
Level of tissue oxygenation and blood volume index of prefrontal and quadriceps muscle tissue | 10 years
  Changes in cerebral and muscle tissue oxygenation will be assessed after 3, 6, 12 months and yearly thereafter by Near-infrared-Spectroscopy
Time, maximal power in stair-ascent test | 10 years
  Changes in performance of stair ascent test will be assessed after 3, 6, 12 months and yearly thereafter
Performance in Sit to stand test | 10 years
  Changes in sit- to stand test will be assessed after 3, 6, 12 months and yearly thereafter
Level of C-reactive protein (CRP) | 10 years
  The change in CRP will be registered at 3, 6, 12 months and yearly thereafter, taken from venous blood sample, measured by immunoassay ('Immulite 2000'; 'DPC'; Los Angeles; USA)
Level of N-terminal brain natriuretic peptide (BNP) | 10 years
  The change in BNP will be registered at 3, 6, 12 months and yearly thereafter, taken from venous blood sample, measured by Roche Modular Systems (Roche; Switzerland)

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Ulrich, MD, Principal Investigator — University Hospital Zurich, Department of Pulmonology
Locations (1):
- University Hospital Zürich, Zurich, Switzerland

REFERENCES:
- [Derived] Saxer S, Lichtblau M, Berlier C, Hasler ED, Schwarz EI, Ulrich S. Physical activity in incident patients with pulmonary arterial and chronic thromboembolic hypertension. Lung. 2019 Oct;197(5):617-625. doi: 10.1007/s00408-019-00248-x. Epub 2019 Jul 1. PMID 31263960